CLINICAL TRIAL: NCT03744351
Title: Analysis of B Cell Differentiation in Multiple Sclerosis
Brief Title: B Cell Differentiation in MS
Acronym: ABCD-SEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC18_8909_ABCD-SEP
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: Follicular helper T cells; B cells; Differentiation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteer (Other): * 45 subjects
  * A single visit
  Interventions: Other: Biological Samples
- Clinically Isolated Syndrome (Other): • 35 subjects
  Interventions: Other: Biological Samples
- Non-MS patients with neurological inflammatory disease (Other): • 30 subjects
  Interventions: Other: Biological Samples
- MS patients (remitting or progressive untreated) (Other): * 30 untreated remittent patients
  * 30 progressive untreated patients
  Interventions: Other: Biological Samples

INTERVENTIONS:
Other: Biological Samples — Venous sampling that is performed solely for the purpose of research. The total blood volume taken is 80 ml maximum (8 tubes of 10 ml).
  Arms: Healthy volunteer
Other: Biological Samples — Eight additional 10 ml tubes of blood and an additional 5 ml CSF tube will be taken from the patient during a sample taken for the patient's usual check-up /follow-up.
  Inpatients will also be offered stool removal.
  Arms: Clinically Isolated Syndrome
Other: Biological Samples — The patient will be taken 8 additional tubes of 10 ml of blood (during a blood test performed for the usual assessment of the patient) and an additional 5 ml of CSF in a sample taken for the assessment of the patient.
  Arms: Non-MS patients with neurological inflammatory disease
Other: Biological Samples — Eight additional 10 ml tubes of blood will be taken from the patient during a sample taken for the patient's usual check-up / follow-up.
  Inpatients will also be offered stool removal
  Arms: MS patients (remitting or progressive untreated)

SUMMARY:
Interventional study with minimal risks and constraints, prospective, monocentric.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the Central Nervous System (CNS) affecting primarily young adults. This disease is the leading cause of non-traumatic disability in this population.

MS has long been considered as a T-cell mediated disease. However, the remarkable efficacy of anti-CD20 monoclonal antibodies in this disease has highlighted the major role of B-lymphocytes in the pathophysiology of this disease.

Despite many advances made recently in understanding the role of B-lymphocytes in the pathophysiology of MS, the precise involvement of plasma cells and their function at different stages of the disease remains unclear. In this project, the investigators plan to analyze the differentiation abilities of circulating B-lymphocytes in patients with MS.

Follicular helper T cells (TFH) play a crucial role in B lymphocyte differentiation. These cells are located within germinal centers in secondary lymphoid organs, and their memory compartment also circulates in the blood. Several circulating TFH subpopulations have recently been defined, with different helping capacities. There is currently very little data on these cells in MS patients. The investigators therefore plan, in a second step, to characterize the phenotype of the different subpopulations of TFH at the periphery, but also in the CSF of MS patients.

ELIGIBILITY:
Inclusion Criteria:

Regarding MS patients (remitting or progressive untreated):

* Adult (age greater than or equal to 18 years) of both sexes;
* MS fulfilling the criteria of McDonald 2017;
* Remittent or progressive form;
* No immunomodulatory or immunosuppressive therapy for at least 3 months;
* Free, informed and written consent signed by the patient.

Regarding Clinically Isolated Syndrome:

* Adult (age greater than or equal to 18 years) of both sexes;
* Clinically isolated syndrome suggestive of MS (at least two typical lesions in two different locations);
* Patient receiving a Lumbar Puncture (PL) for diagnostic purposes;
* No immunomodulatory or immunosuppressive therapy for at least 3 months;
* Free, informed and written consent signed by the patient.

Regarding non-MS patients with neurological inflammatory disease:

* Adult (age greater than or equal to 18 years) of both sexes;
* Patient with non-MS neurological inflammatory disease (examples: meningitis, neurolupus, neurosarcoidosis...);
* Patients with PL for diagnostic or surveillance purposes;
* No immunomodulatory or immunosuppressive therapy for at least 3 months;
* Free, informed and written consent signed by the patient.

Regarding healthy volunteers:

* Adult (age greater than or equal to 18 years) of both sexes;
* Free, informed and written consent signed by the volunteer.

Exclusion Criteria:

Regarding all patients:

* Pregnancy;
* Breastfeeding;
* Treatment with corticotherapy in the last month;
* Patient not affiliated to social security;
* Persons major subject to legal protection (safeguard of justice, guardianship, tutorship), persons deprived of their liberty.

Regarding healthy volunteers:

* Pregnancy;
* Breastfeeding;
* Not affiliated to social security;
* Persons major subject to legal protection (safeguard of justice, guardianship, tutorship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Plasmablasts frequency | At Day 6 after differentiation of B cells
  Frequency of plasmablasts CD38hiCD27hi obtained after 6 days of differentiation of B cells in vitro, analyzed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Laure Michel, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France